CLINICAL TRIAL: NCT05872009
Title: The GaP Study: Gestational Diabetes Mellitus: "Placental-maternal Crosstalk and Future Health
Brief Title: Gestational Diabetes Mellitus: "Placental-maternal Crosstalk and Future Health"
Acronym: GaP
Status: Not yet recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian SIDS and Stillbirth Society (Other)
Responsible Party: Principal Investigator, Meryam Sugulle, Principal Investigator, Oslo University Hospital
Other Study IDs: 494097
Record Dates: First submitted 2023-03-08; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Gestational Diabetes; Cardiovascular Diseases; Placenta Diseases
MeSH Terms: conditions — Diabetes, Gestational; Cardiovascular Diseases; Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood (serum, plasma)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with gestational diabetes: Any treatment. N=200.
- Control group: Gestational-age matched, euglycemic, normotensive pregnant women (n=150)

SUMMARY:
The GaP study is designed to close important knowledge gaps by:

1. exploring placental health and cellular ageing in GDM and the association with neonatal outcome
2. evaluating the effectiveness of current and novel maternal health follow-up strategies after GDM

DETAILED DESCRIPTION:
The incidence of gestational diabetes mellitus (GDM) is increasing. GDM has potential adverse short and long term health effects for both the women and her offspring, and involves dysfunctional interaction between placenta and the maternal body. The burden for the individual, the health system and society warrants further investigations into the placental-maternal crosstalk in GDM in order to improve personalized pregnancy surveillance and follow-up. In Oslo county, nearly twice as many women who give birth suffer from GDM (5.7%) than from preeclampsia (2.3%). The large obstetric department at Ullevål provides an optimal environment for novel translational studies and clinical practical aspects of GDM. The GaP study is designed to close important knowledge gaps by:

1. exploring placental health and cellular ageing in GDM and the association with neonatal outcome
2. evaluating the effectiveness of current and novel maternal health follow-up strategies after GDM

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >18 years with GDM giving birth at Oslo University hospital Ullevål.
* Control group of gestational age matched euglycemic, normotensive pregnancies

Exclusion Criteria:

* reduced fetal movements,
* epilepsy
* thyroidea dysfunction
* hypertensive disorder of pregnancy
* non-communicable disease
* Communicable disease (such as HIV)
* type 1 or type 2 diabetes.
* not able to understand Norwegian or English.
* under legal guardianship.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women with GDM (diagnosed according to guidelines and referred to our outpatient clinic) and healthy, euglycemic pregnant women (Control group: referred for breech evaluation, planning of elective cesarean section, suspected reduced or increased fetal growth with a normal finding at ultrasound). Patients can be recruited from outpatient clinic, prior to induction, at admission for elective cesaerean section or at admission for labor (but not yet in active labor)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of women with altered levels of circulating senescence markers | 4 years
  Levels of maternal circulating senescence markers, e.g. SAA1, free thiol and related markers, in case group compared to controls
Number of women with altered levels of tissue-based senescence markers | 4 years
  Expression of markers of senescence in placental tissue, as assesed by immunohistochemistry (e.g. IL-6, p21, p16 and related markers) in case group compared to controls
Number of women with increased values for postpartum surrogate markers for impaired cardiovascular function | 4 years
  As assessed by circulating maternal levels of cardiovascular biomarkers, e.g. HDL (mmol/l), LDL (mmol/l) and related markers in case group compared to controls
Number of women with increased values for postpartum surrogate markers for impaired cardiovascular function | 4 years
  As assessed by circulating maternal levels of cardiovascular biomarkers, e.g. GDF-15 (ng/l), NT-pro BNP (ng/l), Troponin (ng/l) and related markers in case group compared to controls
Number of neonates with adverse neonatal outcome | 4 years
  A composite measure for neonatal outcome will be created using information on fetal acidemia, Apgar-score, asphyxia, intra-/postpartum fetal death, neonatal intubation/mechanical ventilation, meconium aspiration syndrome, netonatal hypoxic-ishcemic encephalopathy, therapeutic hypothermia of the neonate, rate of acute cesarean section (due to suspected fetal distress) and compared in case group and controls

SECONDARY OUTCOMES:
Number of participants with operative vaginal delivery due to suspected fetal distress | 4 years
  Rates of operative vaginal deliveries (forceps/vacuum/combined; due to suspected fetal distress) in case and control groups
Percentage of participants with pathological placenta histology findings in case and control groups | 4 years
  As assessed by a senior perinatal pathologist using predefined criteria

CONTACTS AND LOCATIONS:
Overall Officials: Meryam Sugulle, PhD, Principal Investigator — Oslo University Hospital, Division of Gynaecology and Obstetrics, Ullevål
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Depending on when the permission for the dataset usage for the project's outcome measures ends (OUH personal data officer/Regional Ethical Comittee) AND Norwegian legislation regarding personal data protection. It is unlikely that a major part of the data set will be shared openly due to these restrictions on sensitive personal data matters.